CLINICAL TRIAL: NCT00525031
Title: Randomized Phase II Neoadjuvant Study of Temozolomide Alone or With Pegylated Interferon-alpha 2b in Patients With Resectable American Joint Committee on Cancer (AJCC) Stage IIIB/IIIC or Stage IV (M1a) Metastatic Melanoma
Brief Title: Temozolomide Alone or With Pegylated Interferon-Alpha 2b (PGI) in Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-0143; NCI-2010-00855 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-08-31; First posted 2007-09-05 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
Keywords: Melanoma; Temozolomide; Temodar; Pegylated Interferon Alpha-2b; PEG-Intron; PGI; Resectable metastatic melanoma; Surgery
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; peginterferon alfa-2b

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temozolomide (TMZ) (Experimental): Temozolomide = TMZ - 150 mg/m^2 by mouth once daily for 7 days, followed by 7 days off (alternating weekly) for a total of 8 weeks.
  Interventions: Drug: Temozolomide (TMZ)
- Temozolomide (TMZ) + Pegylated Interferon-alpha 2b (PGI) (Experimental): Temozolomide = TMZ and PGI = Pegylated Interferon-alpha 2b
  Temozolomide 150 mg/m^2 by mouth once daily for 7 days, followed by 7 days off (alternating weekly) for a total of 8 weeks. Pegylated Interferon-alpha 2b 0.5 mcg/kg subcutaneous injection once weekly for a total of 8 weeks.
  Interventions: Drug: Temozolomide (TMZ); Drug: Pegylated Interferon Alpha-2b (PGI)

INTERVENTIONS:
Drug: Temozolomide (TMZ) — 150 mg/m^2 by mouth once daily for 7 days, followed by 7 days off (alternating weekly) for a total of 8 weeks.
  Other Names: Temodar
Drug: Pegylated Interferon Alpha-2b (PGI) — 0.5 mcg/kg subcutaneous injection once weekly for a total of 8 weeks.
  Other Names: PEG-Intron
  Arms: Temozolomide (TMZ) + Pegylated Interferon-alpha 2b (PGI)

SUMMARY:
The goal of this clinical research study is to learn if temozolomide alone or given with pegylated interferon alpha-2b can help to control metastatic melanoma. Researchers also want to study the safety of these 2 treatments.

Objectives:

1. To determine the anti-tumor activity (pathological response CR+PR) and toxicity of temozolomide (TMZ) alone or in combination with pegylated interferon alpha-2b (PGI) in patients with resectable stage IIIC or stage IV (M1a) metastatic melanoma prior to definitive surgical resection.
2. To determine the relapse-free survival, overall survival and the impact of tumor response to chemotherapy in these patients.
3. To differentiate the in vivo treatment effects of TMZ alone vs.TMZ plus PGI and correlate with clinical outcome by analysis the pre- and post-treatment tumors and peripheral blood mononuclear cells with respect to:

1) Known cellular and molecular markers of apoptosis and cell proliferation, 2) Promotor methylation status of the DNA repair enzyme O6-methylguanine-DNA methyltransferase (MGMT), 3) DNA sequence variability of tumor suppressor genes and DNA repair enzymes, 4) Tumor genomic expression profiles analysis by complementary DNA (cDNA) microarray and protein array

DETAILED DESCRIPTION:
Temozolomide is a drug that is designed to work by stopping cancer cells from making new DNA. If they cannot make DNA, they can't split into 2 new cancer cells.

Pegylated Interferon alpha-2b is a protein made by the human immune system that helps to fight viral infections and regulate cell function.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups (Arm A or Arm B). You have an equal chance of being assigned to either group and getting the treatment assigned to that group. You will not know which group you are assigned to.

Arm A: Participants in this group will take temozolomide once a day for 7 days in a row. This will be followed by 7 days without any treatment. This will be repeated 3 more times(for a total of 8 weeks - 1 cycle) before you have routine surgery.

Arm B: Participants in this group will take temozolomide on the same schedule as those in Arm A. However, participants in this group will also receive pegylated interferon alpha-2b as an injection under the skin once a week for a total of 8 weeks before they have routine surgery. Tylenol will be given to participants in this group before their pegylated interferon alpha-2b injection. After the first injection, they will also need to stay in the clinic for 2 hours of observation.

Your body weight will be used when calculating the dosage of Temozolomide.

You will have blood (about 1 tablespoon each time) drawn at 2 times, to check your response to treatment. The first sample will be drawn before you start treatment. The second sample will be drawn around Day 57 of treatment.

On Days 15, 29, 43, and 57 of treatment, you will be asked about any illness you have experienced and any medications you may be taking. You will have a physical exam, including measurement of vital signs. You will have tumor measurements and a performance status evaluation. You will also have about 1 tablespoon of blood drawn for routine tests at each visit . Any side effects you may have experienced will also be recorded.

All participants will receive 1 cycle (8 weeks) of treatment followed by surgery to remove the tumor. The size of the tumor will be closely monitored during study treatment. If the tumor increases in size by 50% (half) or greater, study treatment will be stopped and you will immediately have surgery. If you have to stop treatment due to side effects from the drug(s), you may be able to start up again once the side effect has gone away or decreased in severity enough. However, the time you are off therapy will count towards the total 8 weeks that you can receive treatment. If recovery from the side effect requires a total of 8 weeks or more from the start of treatment, you will be removed from the study and receive surgery. Tumor and blood samples will be collected during surgery to check how the disease is responding to treatment.

Your routine surgery will be scheduled to take place up to 90 days following completion of your treatment and as soon as your blood counts have recovered to the normal level.

After surgery, if you are experiencing side effects from the study drugs, but show stable disease or you are responding to treatment, you will be able to receive 3 additional cycles of therapy (24 weeks). You will have a physical exam, including measurement of vital signs and routine blood tests (about 1 tablespoon) every 4 weeks. You will then be followed every 3 months with routine blood tests (about 1 tablespoon each time) for the first 3 years, and every 6 months up to 8 years. After that, follow-up will be at the discretion of your primary physician. CT scans of your chest, abdomen, and pelvis will be performed after each cycle of therapy for the 3 additional cycles, then every 6 months up to 5 years and then, at the discretion of your primary physician.

This is an investigational study. Temozolomide alone and given with pegylated interferon alpha-2b is authorized for use in research only. Neither of these drugs is currently approved by the FDA for this treatment. About 124 patients will be enrolled on this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented diagnosis of melanoma metastases.
2. Stage IIIB/IIIC (N2b, N2c and N3) or stage IV (M1a) melanoma patients with measurable and potentially resectable metastases without clinical and radiological evidence of other distant metastases.
3. An Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Age 18 or older.
5. Adequate organ function defined as follows: a.) Absolute granulocytes greater than or equal to 1,000/mm^3 and Platelets greater than or equal to 100,000/mm^3, b.) Serum bilirubin and serum creatinine of less than or equal to 1.5 times upper limit of laboratory normal. If serum creatinine is greater than 1.5 times upper limit of laboratory normal, the urine creatinine clearance must be greater than 60 ml/min., c.) serum glutamate oxaloacetate transaminase (SGOT) (AST), serum glutamate pyruvate transaminase (SGPT) (ALT) and alkaline phosphatase less than or equal to 3 times upper limit of laboratory normal.
6. Patients have not had any previous systemic chemotherapy for metastatic melanoma. Prior biologic therapy, targeted therapy or immunotherapy are allowable, but must be at least 2 weeks since prior therapy before starting study drugs. No other concurrent chemotherapy, immunotherapy, or radiotherapy.
7. Prior radiation therapy used to enhance local regional control is permitted, but must be at least 2 weeks since prior therapy before starting study drugs. In addition, the patient must have unirradiated metastatic sites for response evaluation and has fully recovered from its toxicity. Lesions within the prior field of radiation may only be used as indicator lesions if there has been recent evidence of disease progression after .
8. Ability to understand and sign an informed consent form, indicating awareness of the investigational nature of this study.

Exclusion Criteria:

1. Significant cardiac or pulmonary dysfunction, such as a history of severe cardiovascular disease, myocardial infarction within 6 months of the start of treatment, unstable angina, Class III or Class IV congestive heart failure, ventricular arrhythmia, or any uncontrolled arrhythmia.
2. Current significant psychiatric illness.
3. Serious infection requiring intravenous antibiotics, or any non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by complications of this therapy.
4. Frequent vomiting or any medical condition (e.g. partial bowel obstruction) that could interfere with oral medication intake.
5. Autoimmune or immunosuppressive disorders (e.g. HIV or AIDS-related illness).
6. Patients who require therapy with systemic corticosteroids.
7. No evidence of active secondary malignancy that requires chemotherapy within the past 2 years (excluding non-melanoma skin cancer, and/or all carcinoma in-situ)
8. Pregnant or lactating women are ineligible. Women of childbearing potential must have a negative urine pregnancy test within a week of initiation of therapy. All patients must agree to use medically approved contraceptive measures to prevent pregnancy during treatment.
9. Any other medical condition or reason that, in the principal investigator's opinion, makes the patient unsuitable to participate in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 31, 2006 to May 10, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Three participants of 55 enrolled were excluded due to ineligibility prior to assignment to groups.
Groups:
- Temozolomide (TMZ): TMZ 150 mg/m^2 oral once daily for 7 days, followed by 7 days off (alternating weekly) for a total of 8 weeks.
- Temozolomide (TMZ) + Pegylated Interferon-alpha 2b (PGI): TMZ 150 mg/m^2 oral once daily for 7 days, followed by 7 days off (alternating weekly) and PGI 0.5 mcg/kg subcutaneous injection once weekly for a total of 8 weeks.
Period: Overall Study
Arm/Group | Temozolomide (TMZ) | Temozolomide (TMZ) + Pegylated Interferon-alpha 2b (PGI)
Started | 27 | 25
Completed | 26 | 24
Not Completed | 1 | 1
Not completed — Disease Progression | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- TMZ Alone: TMZ 150 mg/m^2 oral once daily for 7 days, followed by 7 days off (alternating weekly) for a total of 8 weeks.
- TMZ + PGI: TMZ 150 mg/m^2 oral once daily for 7 days, followed by 7 days off (alternating weekly) and PGI 0.5 mcg/kg subcutaneous injection once weekly for a total of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | TMZ Alone | TMZ + PGI | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 71] | 62 [32 to 82] | 60 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 13 | 16 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Response to Neoadjuvant Therapy by Therapy Arms: Clinical Response Rates (CR + PR + SD)
Description: Response to neoadjuvant therapy reported as number of participants with clinical response, defined as Complete Response (CR), Partial Response (PR) or Stable Disease (SD). Clinical Complete Response (CR): Disappearance of all clinical evidence of visible tumor. Partial Response (PR) : 30% or > decrease in the sum of the of the longest diameter of target lesions, taking as reference the baseline sum longest diameter persisting for at least 4 weeks. Progressive Disease (PD): > 20% increase in sum of longest diameter of target lesions, reference baseline sum longest diameter. Appearance new lesions and/or unequivocal progression of existing non-target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, reference smallest sum longest diameter since treatment started.
Time Frame: Evaluated after a total of 8 weeks of therapy before definitive surgery.
Population: Of the 52 registered, two were not evaluable for response. Each
Measure: Count of Participants; unit: Participants
Arm/Group | TMZ Alone | TMZ + PGI
Number analyzed (Participants) | 26 | 24
Participants
  CR, PR, SD | 4 | 7
  PD | 14 | 11
  Missing | 8 | 6

2. Primary Outcome: Response to Neoadjuvant Therapy: Overall Clinical Responses
Description: Response to neoadjuvant therapy reported as number of participants with clinical response, defined as Clinical Complete Response (CR): Disappearance of all clinical evidence of visible tumor. Partial Response (PR) : 30% or > decrease in the sum of the of the longest diameter of target lesions, taking as reference the baseline sum longest diameter persisting for at least 4 weeks. Progressive Disease (PD): > 20% increase in sum of longest diameter of target lesions, reference baseline sum longest diameter. Appearance new lesions and/or unequivocal progression of existing non-target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, reference smallest sum longest diameter since treatment started.
Time Frame: Evaluated after a total of 8 weeks of therapy before definitive surgery.
Population: Two participants of 52 enrolled were not evaluable for response.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Arm A: TMZ 150 mg/m^2 oral once daily for 7 days, followed by 7 days off (alternating weekly) for a total of 8 weeks. Arm B: TMZ 150 mg/m^2 oral once daily for 7 days, followed by 7 days off (alternating weekly) and PGI 0.5 mcg/kg subcutaneous injection once weekly for a total of 8 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Participants
  Complete Response | 1
  Partial Response | 15
  Stable Disease | 3
  Progressive Disease | 31

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from first cycle (8 weeks) of neoadjuvant therapy before undergoing surgical resection and up to 3 additional cycles (24 weeks) following definitive surgery as adjuvant therapy for total of 32 weeks.
Arm/Group | TMZ Alone | TMZ + PGI
Serious Adverse Events (participants affected / at risk) | 0/27 | 8/25
Other Adverse Events (participants affected / at risk) | 26/27 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMZ Alone (N=27) | TMZ + PGI (N=25)
LEUKOCYTES INCREASED/Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPHILS INCREASED (ANC/AGC) (Investigations) | 0 (0) | 1 (1)
LYMPHOPENIA (Investigations) | 0 (0) | 3 (3)
PLATELETS DECREASED (Investigations) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMZ Alone (N=27) | TMZ + PGI (N=25)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
ALANINE TRANSAMINASE (ALT) INCREASED (Investigations) | 0 (0) | 6 (6)
ANOREXIA (Metabolism and nutrition disorders) | 10 (10) | 9 (9)
ASPARTATE AMINOTRANSFERASE (AST) INCREASED (Investigations) | 0 (0) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 11 (11) | 14 (14)
CYSTITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 5 (5)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
ELEVEVATED Serum Glutamic-Oxaloacetic Transaminase (SGOT) (Investigations) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 12 (12) | 17 (17)
FEVER WITHOUT NEUTROPENIA (General disorders) | 0 (0) | 3 (3)
FLU-LIKE SYNDROME (General disorders) | 1 (1) | 7 (7)
HEARTBURN (General disorders) | 0 (0) | 2 (2)
HEMOGLOBIN INCREASED (Investigations) | 3 (3) | 4 (4)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
INDIGESTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INJECTION SITE REACTION (Injury, poisoning and procedural complications) | 1 (1) | 14 (14)
LEUKOCYTES INCREASED/Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 7 (7)
LEUKOPENIA (Investigations) | 2 (2) | 5 (5)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
LYMPHOPENIA (Investigations) | 5 (5) | 7 (7)
MOOD ALTERATION (Psychiatric disorders) | 0 (0) | 3 (3)
NAUSEA (General disorders) | 11 (11) | 16 (16)
NEUTROPHILS DECREASED (Absolute neutrophil count/ANC) (Investigations) | 2 (2) | 7 (7)
PAIN (EXTREMITY-LIMBS) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
PAIN (HEAD/HEADACHE) (Nervous system disorders) | 8 (8) | 16 (16)
PAIN (MUSCLE) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN (SKIN) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PLATELETS DECREASED (Investigations) | 5 (5) | 10 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
RIGORS/CHILLS (General disorders) | 0 (0) | 1 (1)
SWEATING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TASTE ALTERATION (Nervous system disorders) | 1 (1) | 3 (3)
VOMITING (Gastrointestinal disorders) | 4 (4) | 6 (6)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes